CLINICAL TRIAL: NCT01224262
Title: A Randomized, Observer-Blind, Controlled Phase 1/2a Study of the Safety, Tolerability and Immunogenicity of Fluzone Administered With and Without LIQ001 in Two Cohorts of Healthy Subjects: 18-49 Years of Age and 65 Years of Age or Older.
Brief Title: A Study Evaluating the Safety and Tolerability of a Seasonal Influenza Vaccine Containing LIQ001
Acronym: LIfT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: Accelovance (Industry); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LIQC10-001
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: influenza vaccine; seasonal influenza; novel vaccine; flu
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Fluzone + 0.45 mg LIQ001 (Experimental): Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine) Administered with LIQ001 (0.45mg)
  Interventions: Biological: Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine); Biological: LIQ001 (0.45mg)
- Fluzone + 1.8 mg LIQ001 (Experimental): Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine) Administered with LIQ001 (1.8mg)
  Interventions: Biological: Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine); Biological: LIQ001 (1.8mg)
- Fluzone (Active Comparator): Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine)
  Interventions: Biological: Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine)

INTERVENTIONS:
Biological: Fluzone® (2010/2011 Inactivated Trivalent Influenza Vaccine) — A single vaccination of Fluzone alone
  Other Names: seasonal influenza vaccination; seasonal influenza vaccine; seasonal flu vaccination; seasonal flu vaccine
Biological: LIQ001 (0.45mg) — A single vaccination of 0.45 mg LIQ001
  Arms: Fluzone + 0.45 mg LIQ001
Biological: LIQ001 (1.8mg) — A single vaccination of 1.8 mg LIQ001
  Arms: Fluzone + 1.8 mg LIQ001

SUMMARY:
This study is designed to evaluate the safety, tolerability, and immune response of LIQ001 mixed with a commercially available seasonal influenza vaccine (Fluzone) in two populations of subjects; healthy adult subjects 18 to 49 years of age and healthy elderly subjects 65 years of age or older.

DETAILED DESCRIPTION:
Significant advances have been made in the design and delivery of vaccines for the prevention of influenza over the decades. However, two major hurdles remain in the global approach to influenza prevention. First, recent epidemiology research has demonstrated that immune response and protection in elderly populations are suboptimal resulting in significant seasonal influenza disease in this population every year. Second, while preparations for the emergence of pandemic influenza strains have progressed, current egg-based manufacturing methods have not provided sufficient global capacity. Furthermore, the genesis and scale-up of other manufacturing platforms will not rapidly solve this problem. Thus, safe and effective ways are needed to improve protection in the elderly as well as reduce the antigen dose in younger populations in preparation for global needs of pandemic vaccines.

Historically it is known that presentation of antigens in particulate form, for a wide range of pathogens, has clear advantages over the presentation of soluble antigen alone. A novel approach using highly uniform particles has been developed which utilizes size, shape, and composition to control the delivery and presentation of the vaccine antigen(s) to the immune system. Production of these highly uniform particles is possible because of a proprietary manufacturing approach called Pattern Replication in Non-wetting Templates (PRINT®).

The proposed approach is to use the PRINT process to make bioabsorbable particles to improve the immune response and efficacy of the seasonal influenza vaccine. It is proposed that mixing properly sized and charged particles with commercial trivalent influenza vaccine (TIV) will increase vaccine effectiveness and/or decrease the amount of antigen necessary to induce an immune response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 49 years (Cohort 1) and age 65 or above (Cohort 2)
* For subjects 18 to 49 years of age: in good health as determined by medical history, physical examination, and the clinical judgment of the Principal Investigator (PI)
* For subjects 65 years of age and older: in stable good health as determined by medical history, physical examination, and the clinical judgment of the PI
* Live in the community (including assisted living)
* Available for duration of study (1 year)
* If female, no child-bearing potential or using appropriate measures to prevent pregnancy
* Negative urine pregnancy test for women presumed to be of child-bearing potential within 24 hours of vaccination
* Be eligible for screening
* Provide informed consent
* Have working phone for contact by the study site personnel

Exclusion Criteria:

* Known allergy to eggs or any other component of Fluzone (including natural latex) or inactivated influenza vaccines or the investigational vaccine
* Received seasonal influenza or H1N1 vaccine in last 6 months
* A diagnosis of influenza within the previous 12 months
* Received any licensed vaccine within the past 1 month
* Receiving nursing home or equivalent care
* For women, breast-feeding or planning to become pregnant during the first three months post-vaccination
* Chronic administration of immunosuppressant(s) or other medication that modifies immune function
* Confirmed immunodeficiency syndrome or disease
* Significant cardiovascular disease including class 3 or 4 congestive heart failure, recent history (last 6 months) of acute myocardial infarction, coronary artery bypass surgery or stent placement, unstable angina, uncontrolled arrhythmia, and for subjects 65 years of age and older, a resting heart rate greater than 100 bpm
* Hypertension that is not well controlled by medication in the judgment of the investigator or is more than 150/95 at enrollment
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Medically significant chronic lung disease, e.g., requiring chronic steroid treatment (oral doses >10 mg/day)
* Asthma that is severe, unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral, intravenous, or high dose inhaled corticosteroids (mild or intermittent asthma treated with inhaled steroids is acceptable)
* Medically significant acute or progressive hepatic disease
* Medically significant acute or progressive renal disease
* Diabetes mellitus type 2 not under pharmacological control
* A diagnosis of cancer with active treatment within the previous 5 years (except for a localized basal cell carcinoma of the skin)
* History of autoimmune/inflammatory conditions (e.g., rheumatoid arthritis and diabetes mellitus type 1)
* Medically significant acute or progressive neurological disease.
* Seizure disorder that has required treatment within the last 3 years
* History of Guillain-Barre Syndrome (GBS)
* Administration of blood products, immunoglobulin, or investigational vaccine in the 3 months prior to immunization in this study
* Use of investigational product (other than blood, immunoglobulin, or vaccine) in the past 60 days
* Seropositive for HCV, HIV or positive for HBsAg
* History of excessive alcohol use, drug abuse, or significant psychiatric illness
* Unable to complete informed consent
* Abnormal laboratory assessment meeting criteria for a mild, moderate, or severe adverse event
* Any other condition or circumstance which, in the opinion of the PI, poses an unacceptable risk for participation in the study
* Inability to operate and answer a telephone and lack of access to telephone
* Temporary Exclusion Criteria: Presence of an oral temperature ≥99.5°F, and/or signs and symptoms of an acute infectious respiratory illness within 3 days prior to vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The rate of Adverse Events attributable to each of the doses of LIQ001 mixed with Fluzone compared to Fluzone alone. | 35 days post-vaccination

SECONDARY OUTCOMES:
HAI response (Geometric Mean Titer) of each of the doses of LIQ001 mixed with Fluzone compared to the Fluzone alone response. | 21 days post-vaccination
HAI response (Percent with HAI titer greater than or equal to 1:40) of each of the doses of LIQ001 mixed with Fluzone compared to the Fluzone alone response. | 21 days post-vaccination
HAI response (Seroconversion rate) of each of the doses of LIQ001 mixed with Fluzone compared to the Fluzone alone response. | 21 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Frank Malinoski, MD, PhD, Study Director — Liquidia Technologies, Inc.
Locations (1):
- Accelovance - Melbourne, Melbourne, Florida, United States